CLINICAL TRIAL: NCT00688883
Title: A Multicenter, Open Study to Assess the Antitumor Effect and Safety of Oral Fludarabine Phosphate (Fludara (SH T 586): 40 mg/m2/Day) Administered in 3 - 6 Treatment Cycles (1 Treatment Cycle: 5-consecutive Day Dosing, Followed by a Observation Period of 23 Days) in Patients With Indolent Lymphoma
Brief Title: Fludara (Oral) Phase II Study for Indolent Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 305621; 91101
Record Dates: First submitted 2008-05-30; First posted 2008-06-03 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Lymphoma
Keywords: Fludarabine; Purine analog; Indolent lymphoma
MeSH Terms: conditions — Lymphoma | interventions — fludarabine phosphate

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Fludarabine Phosphate (Fludara)

INTERVENTIONS:
Drug: Fludarabine Phosphate (Fludara) — Patients received Fludarabine Phosphate orally for 5 consecutive days, followed by a 23-day observation period. Setting this as 1 treatment cycle, 6 cycles will be given.
  Other Names: BAY86-4864

SUMMARY:
To assess the antitumor effect and safety of Fludara in patients with indolent lymphoma.

DETAILED DESCRIPTION:
As of 29 May 2009, the clinical trial sponsor is Genzyme Corporation. NOTE: This study was originally posted by sponsor Schering AG, Germany, which was subsequently renamed to Bayer Schering Pharma AG, Germany.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed indolent lymphoma (including mantle cell lymphoma)
* Patients with measurable lesions (major axis > 1.5 cm by CT)
* Patients who failed to have PR to previous chemotherapies or antibody therapies. Patients with subsequent relapse after a previously attained CR or with subsequent recurrence after a previously attained PR
* Patients who have not received chemotherapies, antibody therapies or radiotherapies for more than 4 weeks (more than 3 months in the case of the antibody therapies)
* Patients who have PS Grade 0 to 2 in the criteria of ECOG
* Patients with adequately maintained organ functions

Exclusion Criteria:

* Patients with infectious disease, serious complications, serious gastrointestinal symptoms, serious bleeding tendency (DIC), CNS metastases, fever more than 38 degrees Celsius, interstitial pneumonia or pulmonary fibrosis, active other malignancies, AIHA or the history of allergies to similar purine analogs
* Patients who are positive for HBs antigen, HCV antibody or HIV antibody
* Patients who received G-CSF or blood transfusion within 1 week before the screening test
* Patients who had ever received previous therapy with fludarabine phosphate injection (Fludara), pentostatin (Coforin), cladribine (Leustatin) or SH T 586
* Patients who are pregnant, of childbearing potential, lactating, or who do not agree to practice contraception

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2003-02; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Best overall response rate; Antitumor effect | at screening and re-evaluation, at 4th week or at the time of discontinuation of treatment cycles 1, 3 and 6, and at 12th week after last observation of last treatment cycle

SECONDARY OUTCOMES:
CR rate | after last observation of last treatment cycle
Time to treatment failure | after last observation of last treatment cycle
Overall survival | after last observation of last treatment cycle
Adverse events collection | after last observation of last treatment cycle

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (15):
- Japan (15):
  - Nagoya, Aichi-ken
  - Kashiwa-shi, Chiba
  - Fukuoka, Fukuoka
  - Sapporo, Hokkaido
  - Akashi-shi, Hyōgo
  - Kagoshima, Kagoshima-ken
  - Isehara-shi, Kanagawa
  - Kyoto, Kyoto
  - Sendai, Miyagi
  - Nagasaki, Nagasaki
  - Okayama, Okayama-ken
  - Moriguchi-shi, Osaka
  - Hamamatsu, Shizuoka
  - Chuo-ku, Tokyo
  - Shinjuku-ku, Tokyo